CLINICAL TRIAL: NCT03149133
Title: Comparison of Occlusive and Classical Hypertrophy Training in Terms of Thickness and Stiffness of The Muscle, An Ultrasound-Based Study
Brief Title: Comparison of Occlusive and Classical Hypertrophy Training in Terms of Thickness and Stiffness of The Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, ÖMER BATIN GÖZÜBÜYÜK, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2016/248
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Muscle Tightness; Hypertrophy; Occlusion Vein
Keywords: Biomechanics; Strength training; Elastography; Ultrasound
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor are blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Hypertrophy (Experimental): The classical hypertrophy group performs strength training with 75-80% of 1-Repetition Maximum.
  Interventions: Other: Heavy hypertrophy training
- Occlusive Training (Experimental): The occlusive hypertrophy group performs strength training with %35-50 of 1-Repetition Maximum.
  Interventions: Other: Light hypertrophy training

INTERVENTIONS:
Other: Heavy hypertrophy training — Training with 75-80 % of 1-RM
  Arms: Classical Hypertrophy
Other: Light hypertrophy training — Training with 35-50 % of 1-RM
  Arms: Occlusive Training

SUMMARY:
Occlusive or ischemic training is a type of strength training which is becoming more and more popular every day. The safety, efficacy and detailed description about the use of occlusive training is well documented in the literature. However, the effects on hypertrophy and the stiffness of the muscle tissue are not studied. We aimed to measure these changes by ultrasound technology in a randomized controlled design.

DETAILED DESCRIPTION:
Patients were randomized into classical hypertrophy and occlusive hypertrophy groups. The participants are free from any systemic disease, infection or recent injury. Both groups perform hypertrophy training with different intensities. The outcome measures are; thickness determined by B-mode ultrasound and stiffness by shear-wave elastography. Comparison of both groups will be made.

ELIGIBILITY:
Inclusion Criteria:

* Healthy recreational athletes

Exclusion Criteria:

* Any kind of systemic disorder
* Active or chronic infection
* Recent (last 6 months) musculoskeletal injury
* Performed strength training at last 72 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Thickness | 6 weeks
  The thickness of the biceps brachii muscle determined by B-mode ultrasound
Stiffness | 6 weeks
  The stiffness of the biceps brachii muscle determined by ultrasound elastography

SECONDARY OUTCOMES:
Strength change | 6 weeks
  Arm flexion strength determined by isokinetic dynammometer

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided